CLINICAL TRIAL: NCT05270330
Title: The Relationship Between Plaque Stability Evaluated by IVUS and Metabolomics in Stable Coronary Heart Disease Patients
Brief Title: Plaque Stability and Metabolomics in Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaanxi Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhongwei, Professor, Shaanxi Provincial People's Hospital
Other Study IDs: 2021BJ-02
Record Dates: First submitted 2022-01-22; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
Keywords: plaque stability; metabonomics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is an observational study, we don't have any interventions. — No intervention

SUMMARY:
At present, the investigators don't know the relationship between plaque stability and the metabonomics changes. In the present study, investigators will evaluate the plaque stability by intravascular unltrasound in stable coronary heart patients, and metabonomics was also assessed by high throughput sequencing. Statistic analysis were carried out to analyze the correlation between plaque stability and metabonomics changes among these study patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed with stable coronary heart disease and evaluated for plaque stability by IVUS will be recruited.

Exclusion Criteria:

* renal insufficiency with serum creatinine > 20 mg/L;
* regnant/lactating women, or the women receive hormone replacement therapy in premenopausal or postmenopausal;
* patients have a history of abusing alcohol or other drugs in the past two years, active hepatitis, cirrhosis;
* endocrine abnormalities without therapy (diabetic ketoacidosis, thyroid disease, etc.);
* The body's inflammatory disease, rheumatoid arthritis, osteoarthritis, ulcerative bowel disease, systemic lupus erythematosus (sle), etc.), myositis/myopathy, cancer;
* Dilated cardiomyopathy, valvular heart disease, persistent atrial fibrillation;
* patients recently injured;（8）Other researchers don't agree to join this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with stable coronary heart disease and assessed for plaque stability by IVUS will be recruited in our study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Plaque stability | 07/01/2021-07/31/2024
  The investigators will use the intravascular ultrasound to assess the coronary plaque stability of the patients with coronary heart disease.

SECONDARY OUTCOMES:
Metabonomics | 07/01/2021-07/31/2024
  Serum or plasma will be collected by the investigators and high-throughput sequencing will be used to assess the metabonomics of patients with coronary heart disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaanxi Provincial People's Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No